CLINICAL TRIAL: NCT05805215
Title: Noninvasive Temporal Interference Stimulation: An Approach for Modulating Associative Memory by Targeting Deep-brain Targets
Brief Title: Noninvasive Temporal Interference Stimulation: Modulating Associative Memory by Targeting Deep-brain Targets
Acronym: Deep-HiPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LX22NPO5107
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy Aging; Memory Disorders in Old Age; Mild Cognitive Impairment; Alzheimer Disease
Keywords: temporal interference stimulation; associative memory; hippocampus; precuneus; fMRI; EEG
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will undergo 3 types of TIS in randomized order:
  1. targeting the hippocampus
  2. targeting the precuneus
  3. control condition with high-frequency stimulation
Who Masked: Participant, Care Provider
Masking Description: The study participant and researcher applying brain stimulation will be blinded to the stimulation condition. high-frequency stimulation (>1Khz) will be used as a control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active TIS of the hippocampus (Experimental): Participants will undergo Active TIS of the hippocampus as one of the 3 conditions within the trial in randomized order.
  Interventions: Combination Product: Non-invasive Temporal Interference stimulation and Face-name association training task targeting the hippocampus
- Active TIS of the precuneus (Experimental): Participants will undergo Active TIS of the precuneus as one of the 3 conditions within the trial in randomized order.
  Interventions: Combination Product: Non-invasive Temporal Interference stimulation and Face-name association training task targeting the Precuneus
- High-frequency stimulation (Placebo Comparator): High frequency >1Khz stimulation; Assumption: The intrinsic low-pass filtering of electrical signals by the neural membrane prevents neural electrical activity from following very high-frequency oscillating (e.g., > 1 kHz) electric fields.
  Interventions: Combination Product: High-frequency stimulation (placebo) with Face-name association training task

INTERVENTIONS:
Combination Product: Non-invasive Temporal Interference stimulation and Face-name association training task targeting the hippocampus — TIS relies on high frequencies which can penetrate with relatively low loss. High-frequency carriers (>1 kHz) emitted by two (or more) pairs of cutaneous electrodes can temporally interfere at deep peripheral nerve targets. The effective stimulation frequency is equal to the offset frequency between the carriers. By controlling field orientation and frequency offset, the hot spot of constructive interference can be precisely targeted. The key aspect of this method is the use of carrier waves at frequencies higher than 1 kHz. Frequencies above this range are regarded as non-stimulating and pass-through tissues with relatively low loss. While these higher frequencies do not stimulate neural tissue, the interference envelope of two phase-shifted frequencies can elicit action potentials because the offset (aka "beat") frequency can be tuned accordingly to < 100 Hz.
  Arms: Active TIS of the hippocampus
Combination Product: Non-invasive Temporal Interference stimulation and Face-name association training task targeting the Precuneus — TIS relies on high frequencies which can penetrate with relatively low loss. High-frequency carriers (>1 kHz) emitted by two (or more) pairs of cutaneous electrodes can temporally interfere at deep peripheral nerve targets. The effective stimulation frequency is equal to the offset frequency between the carriers. By controlling field orientation and frequency offset, the hot spot of constructive interference can be precisely targeted. The key aspect of this method is the use of carrier waves at frequencies higher than 1 kHz. Frequencies above this range are regarded as non-stimulating and pass-through tissues with relatively low loss. While these higher frequencies do not stimulate neural tissue, the interference envelope of two phase-shifted frequencies can elicit action potentials because the offset (aka "beat") frequency can be tuned accordingly to < 100 Hz.
  Arms: Active TIS of the precuneus
Combination Product: High-frequency stimulation (placebo) with Face-name association training task — High-frequency (>1 kHz) stimulation; Standardly used as a carrier frequency; Effects are expected to he high-pass filtered by neurons
  Arms: High-frequency stimulation

SUMMARY:
Alzheimer's disease and its preclinical stages are characterized by progressive neurodegenerative changes in the hippocampi and default mode network resulting in dysfunctions in episodic memory and its central part the associative memory. Associative memory allows for learning and remembering the relationship between unrelated items. Previous research suggests that non-invasive brain stimulation can influence associative memory but with the caveat of quite a small precision and relatively small effects due to the ability only influence superficial brain areas. Novel Brain stimulation techniques such as temporal interference stimulation (TIS) allow overcoming these caveats by allowing focal non-invasive deep brain stimulation. The main goal of this pilot clinical trial is to modulate associative memory among healthy seniors by influencing the cortico-hippocampal circuits using TIS. Secondly, the goal is to use functional magnetic resonance imaging (fMRI) and EEG to explore the neural correlates of TIS effects on brain networks and find biomarkers that allow predicting better response to brain stimulation.

DETAILED DESCRIPTION:
Alzheimer's disease and its preclinical stages are characterized by progressive neurodegenerative changes in the hippocampi and default mode network resulting in dysfunctions in episodic memory and its central part the associative memory. Encoding of associative information occurs in the distributed brain networks involving the inferior frontal cortex, fusiform cortex, medial temporal lobe, premotor and posterior parietal cortex including the precuneus. Previous studies have shown that by targeting specific nodes within the cortico-hippocampal circuits via the tools of non-invasive brain stimulation the associative memory (AM) performance can be manipulated, however, only relatively surface areas of this circuit were accessible by current non-invasive stimulation techniques. Novel modalities of non-invasive transcranial electrical stimulation such as temporal interference stimulation (TIS) holds a promise to stimulate deeper brain structures without compromising the focality.

TIS relies on high frequencies which can penetrate with relatively low loss. High-frequency carriers (>1 kHz) emitted by two (or more) pairs of cutaneous electrodes can temporally interfere at deep peripheral nerve targets. The effective stimulation frequency is equal to the offset frequency between the carriers. By controlling field orientation and frequency offset, the hot spot of constructive interference can be precisely targeted. The key aspect of this method is the use of carrier waves at frequencies higher than 1 kHz. Frequencies above this range are regarded as non-stimulating and pass-through tissues with relatively low loss. While these higher frequencies do not stimulate neural tissue, the interference envelope of two phase-shifted frequencies can elicit action potentials because the offset (aka "beat") frequency can be tuned accordingly to < 100 Hz. The latest studies showed positive behavioral effects of TIS applied over the primary motor cortex or motor striatum in healthy young adults. To date, no studies have investigated the effect of TIS on AM.

The specific objectives include: 1) Implement a novel temporal interference stimulation (TIS) technique in a proof-of-concept study targeting deep structures of the cortico-hippocampal circuit, which were until this date unattainable reliably by non-invasive stimulation techniques, with the aim to modulate associative memory in healthy seniors. 2) Explore neural underpinnings of TIS effects and find biomarkers associated with better temporal interference stimulation outcomes and with optimal candidates' selection by using EEG/fMRI techniques

ELIGIBILITY:
Inclusion Criteria:

* Intact cognition
* with the ability to comprehend the experimental task
* right-handed

Exclusion Criteria:

* left-handed
* severe internal disease, cancer
* brain tumour, intracranial surgery, psychiatric disorder
* severe neurological brain disease; i.e.: epilepsy, stroke etc.
* the presence of a pacemaker/defibrillator, metal incompatible with magnetic resonance in the body
* incapacitating musculoskeletal disorders
* cognitive impairment based on screening tests
* severe impairment of vision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy in Face-Name association task | Measured during stimulation procedure; assessed through study completion, an average of 2 years
  The face-name association task will be composed of blocks of encoding and recall. Each block contained a unique face-name pair. Multiple pairs followed by a delay and a recall period, where participants tried to select the correct name of each face out of five options (i.e., one target name, two foil names that were present in the block but associated with a different face, and two distracting names that were not present during the task). After each name selection, participants were asked to rate their choice confidence (1, not confident at all to 4, extremely confident)
Speed in Face-Name association task | Measured during stimulation procedure; assessed through study completion, an average of 2 years
  The face-name association task will be composed of blocks of encoding and recall. Each block contained a unique face-name pair. Multiple pairs followed by a delay and a recall period, where participants tried to select the correct name of each face out of five options (i.e., one target name, two foil names that were present in the block but associated with a different face, and two distracting names that were not present during the task). After each name selection, participants were asked to rate their choice confidence (1, not confident at all to 4, extremely confident)

SECONDARY OUTCOMES:
changes in resting-state functional connectivity in regions of interest | Baseline measurement approximately 20 minutes prior stimulation; immediately after stimulation protocol up to 30 minutes
  resting-state fMRI: the analysis will be primarily focused on alterations within nodes in the Default mode Network and between network connectivity; Secondary focus on task-positive networks, namely: Central executive network and Dorsal attentional network
Transcranial magnetic stimulation evoked activity change over the regions of interest (Precuneus, prefrontal cortex) | Baseline measurement approximately 30 minutes prior stimulation; immediately after stimulation protocol up to 40 minutes
  Transcranial magnetic stimulation (TMS) evoked potentials; Investigation of local cortical circuits and networks activated following stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- CEITEC Masaryk university, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salami A, Pudas S, Nyberg L. Elevated hippocampal resting-state connectivity underlies deficient neurocognitive function in aging. Proc Natl Acad Sci U S A. 2014 Dec 9;111(49):17654-9. doi: 10.1073/pnas.1410233111. Epub 2014 Nov 24. PMID 25422457
- [Background] Preston AR, Eichenbaum H. Interplay of hippocampus and prefrontal cortex in memory. Curr Biol. 2013 Sep 9;23(17):R764-73. doi: 10.1016/j.cub.2013.05.041. PMID 24028960
- [Background] Eichenbaum H. Prefrontal-hippocampal interactions in episodic memory. Nat Rev Neurosci. 2017 Sep;18(9):547-558. doi: 10.1038/nrn.2017.74. Epub 2017 Jun 29. PMID 28655882
- [Background] Wagner AD, Shannon BJ, Kahn I, Buckner RL. Parietal lobe contributions to episodic memory retrieval. Trends Cogn Sci. 2005 Sep;9(9):445-53. doi: 10.1016/j.tics.2005.07.001. PMID 16054861
- [Background] Koch G, Bonni S, Pellicciari MC, Casula EP, Mancini M, Esposito R, Ponzo V, Picazio S, Di Lorenzo F, Serra L, Motta C, Maiella M, Marra C, Cercignani M, Martorana A, Caltagirone C, Bozzali M. Transcranial magnetic stimulation of the precuneus enhances memory and neural activity in prodromal Alzheimer's disease. Neuroimage. 2018 Apr 1;169:302-311. doi: 10.1016/j.neuroimage.2017.12.048. Epub 2017 Dec 19. PMID 29277405
- [Background] Lang S, Gan LS, Alrazi T, Monchi O. Theta band high definition transcranial alternating current stimulation, but not transcranial direct current stimulation, improves associative memory performance. Sci Rep. 2019 Jun 12;9(1):8562. doi: 10.1038/s41598-019-44680-8. PMID 31189985
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Background] Wang H, Jin J, Cui D, Wang X, Li Y, Liu Z, Yin T. Cortico-Hippocampal Brain Connectivity-Guided Repetitive Transcranial Magnetic Stimulation Enhances Face-Cued Word-Based Associative Memory in the Short Term. Front Hum Neurosci. 2020 Oct 30;14:541791. doi: 10.3389/fnhum.2020.541791. eCollection 2020. PMID 33192388
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- See also: Related Info — https://www.fnusa-icrc.org/en/npo-project-coordinated-by-fnusa-approved/